CLINICAL TRIAL: NCT05355714
Title: A Single Center, Blinded, Split-Body, Randomized Clinical Trial of High Intensity Ultrasound for the Treatment of Upper Inner Arm Skin Laxity
Brief Title: High Intensity Ultrasound for the Treatment of Upper Inner Arm Skin Laxity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sofwave-Ultherapy-2021-12
Record Dates: First submitted 2022-04-06; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: Treatments will be split-body with subjects receiving treatment from one device on their right side and one on their left.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sofwave (Experimental)
  Interventions: Device: Sofwave
- Ultherapy (Other)
  Interventions: Device: Ultherapy

INTERVENTIONS:
Device: Sofwave — High-Frequency Non-Focused Ultrasound Device
  Arms: Sofwave
Device: Ultherapy — Microfocused Ultrasound with Visualization
  Arms: Ultherapy

SUMMARY:
Upper inner arms of enrolled subjects will be randomized to two (2) treatment groups: Sofwave and Ultherapy, with subjects receiving treatment with one device on their right side and the other on their left.

DETAILED DESCRIPTION:
This is a prospective, single-center, blinded, split-body site, randomized, controlled clinical trial. The study will consist of 15 subjects who will be treated with Sofwave® on one upper medial arm and Ultherapy® to the contralateral upper medial arm for treatment of skin laxity.

Upon enrollment and after a thorough review of the inclusion and exclusion criteria as well as obtaining written and informed consent, each subject will be randomized to have either their right upper inner arm or left upper inner arm treated with Sofwave®, and the contralateral arm will be treated with Ultherapy®. The treatment area is defined as the upper inner medial arm (Appendix A). This area, which abuts the axilla, was chosen as the treatment zone because it is primarily composed of skin on superficial fascia without excessive amounts of adipose tissue. Conversely, the posterior arm typically has extra adipose tissue which would confound the study's measurements

At every visit, the subject's medical history and concomitant medications will be reviewed in detail and weight will be recorded. Additionally, at every treatment and follow-up visit, each subject will have standardized, high-resolution digital photographs taken (Appendix D). Prior to the treatment and at all follow-up visits, the blinded investigator will complete the Upper Inner Arm Visual Crepiness/Laxity Grading Scale, Point of Maximal Upper Arm Skin Laxity Diameter and Circumference Measurements, and skin firmness and elasticity measurements using a Cutometer® Dual MPA 580 (Courage+Khazaka electronic GmbH; Köln, Germany).

Subjects may be treated on the same day that they are screened and provide informed consent. If applicable, a urine pregnancy test will be obtained prior to each treatment. Anesthesia will be provided per physician discretion; options include topical anesthetic (23% lidocaine/7% tetracaine) for 1-hour, oral valium, and/or nitrous oxide. Immediately before treatment, the upper arm treatment zones should be mapped and subsequently cleansed with Hibiclens® (chlorhexidine gluconate solution 4%; Mölnlycke Health Care AB; Gothenburg, Sweden). The arm randomized to receive Sofwave® will receive one treatment session during which the treatment area will receive 3-4 passes. The arm randomized to receive Ultherapy® will receive one treatment session during which the treatment area will receive 1 pass with the 4.0 MHz, 4.5-mm-depth transducer and a subsequent pass with the 7.0 MHz, 3.0-mm-depth transducer. Treatment start and end times will be recorded.

After each treatment session and during all follow-up visits, the treating physician will evaluate the subjects for any procedure-related side effects and adverse events. The subjects will rate their pain. At each follow-up visit, a Physician Global Aesthetic Improvement Scale (PGAIS), Subject Global Aesthetic Improvement Scale (SGAIS), and subject satisfaction questionnaire will be completed.

ELIGIBILITY:
Inclusion Criteria:

a) Male or female subjects > 35 years of age and < 70 years of age b) Subjects in good general health based on investigator's judgment and medical history c) Upper inner arm skin laxity that improves when the skin of the upper inner arm is stretched or lifted superiorly d) Moderate to severe upper inner arm skin crepiness/laxity based on the Upper Inner Arm Visual Crepiness/Laxity Grading Scale (Appendix B) e) Must be willing to give and sign an informed consent form and photographic release form f) Must have a stable body weight for at least six (6) months prior to study entry g) Must be willing to maintain usual sun exposure, diet, and exercise routines for the duration of the study h) Must agree to avoid tanning or use of sunless tanner during the entire course of the study i) Negative urine pregnancy test result at the time of study entry (if applicable) j) For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

1. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
2. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.

k) Must be willing to comply with study treatments and complete the entire course of the study

Exclusion Criteria:

1. Liposuction to bilateral upper arms during the 12-month period prior to study treatment or any time during the course of the study
2. Mesotherapy; dermal fillers, biostimulatory injectables; radiofrequency device treatments; microfocused ultrasound device treatments; laser and light-based device treatments; microneedling; cryolipolysis; high intensity focused electromagnetic energy device treatment; or surgery (i.e., brachyplasty) during the 12-month period before study treatment
3. Any investigational treatment of skin crepiness/laxity of the upper arms during the 12-month period before the study treatment
4. Creams/cosmeceuticals and/or home therapies to prevent or treat skin laxity during the four-week period before study treatment
5. Subjects with scarring in the treatment areas
6. History of thrombosis, post-thrombosis syndrome, or any vascular disorder of the bilateral upper extremities
7. Any history of bleeding or coagulation disorders
8. Subjects with tattoos or permanent implants in the treatment areas
9. Subjects with a significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study
10. Subjects with a history of or presence of any skin condition/disease (including but not limited to any visible rash, atopic dermatitis, psoriasis, actinic keratoses, keratinocyte carcinoma, melanoma, etc.) in the treatment area that might interfere with the diagnosis or evaluation of study parameters
11. Subjects with an active bacterial, viral, or fungal infection of the treatment areas
12. Subjects who spray tanned or used sunless tanners in the treatment areas four (4) weeks prior to study treatment
13. History of lidocaine sensitivity deemed by the investigator to preclude the subject from enrolling into the study
14. Subjects planning any cosmetic procedure to the treatment areas during the study period, other than the treatment that will be performed by the investigator
15. Presence of incompletely healed wound(s) in the treatment area
16. Subject who is on an immunosuppressant or has an autoimmune condition
17. Female subjects who are pregnant, planning a pregnancy, or breast feeding during the study
18. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Upper Inner Arm Visual Skin Crepiness and Laxity | Screening to One Month Post-Treatment
  Upper Inner Arm Visual Skin Crepiness/Laxity Grading Scale completed by blinded investigator
Upper Inner Arm Visual Skin Crepiness and Laxity | Screening to Three Months Post-Treatment
  Upper Inner Arm Visual Skin Crepiness/Laxity Grading Scale completed by blinded investigator
Upper Arm Circumference | Screening to One Month Post-Treatment
  Blinded Investigator Measurement of Point of Maximal Upper Arm Skin Laxity and Circumference
Upper Arm Circumference | Screening to Three Months Post-Treatment
  Blinded Investigator Measurement of Point of Maximal Upper Arm Skin Laxity and Circumference
Upper Arm Firmness | Screening to One Month Post-Treatment
  Blinded Investigator Measurement of Skin Firmness
Upper Arm Firmness | Screening to Three Months Post-Treatment
  Blinded Investigator Measurement of Skin Firmness
Upper Arm Elasticity | Screening to One Month Post-Treatment
  Blinded Investigator Measurement of Skin Elasticity
Upper Arm Elasticity | Screening to Three Months Post-Treatment
  Blinded Investigator Measurement of Skin Elasticity
Physician Global Aesthetic Improvement Scale (PGAIS) | One Month Post-Treatment
  Assessment of overall change in treatment area by blinded investigator
Physician Global Aesthetic Improvement Scale (PGAIS) | Three Months Post-Treatment
  Assessment of overall change in treatment area by blinded investigator

SECONDARY OUTCOMES:
Subject Global Aesthetic Improvement Scale (SGAIS) | One Month Post-Treatment
  Assessment of overall change in treatment area by subject
Subject Global Aesthetic Improvement Scale (SGAIS) | Three Months Post-Treatment
  Assessment of overall change in treatment area by subject
Subject Satisfaction Questionnaire | One Month Post-Treatment
  Subject degree of satisfaction with results of treatment
Subject Satisfaction Questionnaire | Three Months Post-Treatment
  Subject degree of satisfaction with results of treatment
Subject Pain Score | Day of Treatment
  Subject Assessment of Pain During Treatment
Erythema | Day of Treatment
  Treating Investigator Evaluation of Erythema
Erythema | One Month Post-Treatment
  Treating Investigator Evaluation of Erythema
Erythema | Three Months Post-Treatment
  Treating Investigator Evaluation of Erythema
Edema | Day of Treatment
  Treating Investigator Evaluation of Edema
Edema | One Month Post-Treatment
  Treating Investigator Evaluation of Edema
Edema | Three Months Post-Treatment
  Treating Investigator Evaluation of Edema
Dyspigmentation | Day of Treatment
  Treating Investigator Evaluation of Dyspigmentation
Dyspigmentation | One Month Post-Treatment
  Treating Investigator Evaluation of Dyspigmentation
Dyspigmentation | Three Months Post-Treatment
  Treating Investigator Evaluation of Dyspigmentation
Ulceration | Day of Treatment
  Treating Investigator Evaluation of Ulceration/Erosion
Ulceration | One Month Post-Treatment
  Treating Investigator Evaluation of Ulceration/Erosion
Ulceration | Three Months Post-Treatment
  Treating Investigator Evaluation of Ulceration/Erosion

CONTACTS AND LOCATIONS:
Locations (1):
- Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No